CLINICAL TRIAL: NCT02819336
Title: Effectiveness and Safety of Electroacupuncture on Poststroke Urinary Incontinence: a Pilot Multicentered, Randomized, Parallel, Sham-controlled Trial
Brief Title: Effectiveness and Safety of Electroacupuncture on Poststroke Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University (Other)
Collaborators: Wonkwang University Gwangju Medical Center (Unknown)
Responsible Party: Principal Investigator, Lee Eui-ju, Professor, Kyunghee University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016006; KOMCIRB-160215-HR-006 (Other: IRB of Kyung Hee University Korean Medicine Hospital)
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Urinary Incontinence; Stroke, Complication
Keywords: urinary incontinence; electroacupuncture; stroke; complications; randomized controlled trial; pilot projects
MeSH Terms: conditions — Urinary Incontinence; Stroke | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electroacupuncture (EA) group (Experimental): 1. Electroacupuncture therapy (10 sessions within 21 days)
  2. CV2, CV3, CV4, CV6, and bilateral points of SP11, SP6 (8 acupoints in total)
  3. 20 minutes duration with middle frequency (30 Hz) of electrical stimulation
  4. Conventional treatments (drugs, traditional herbal medications, rehabilitation therapies, or acupuncture therapies without electrostimulation for stroke and urinary incontinence / electroacupuncture therapies other than the acupoints (CV2, CV3, CV4, CV6, SP1 and SP6) for stroke and urinary incontinence) are permitted.
  Interventions: Device: Electroacupuncture (EA)
- Park sham (PS) group (Sham Comparator): 1. Non-penetrating Park sham electroacupuncture treatment (10 sessions within 21 days)
  2. CV2, CV3, CV4, CV6, and bilateral points of SP11, SP6 (8 acupoints in total)
  3. 20 minutes duration with undelivered electrostimulation of middle frequency (30 Hz)
  4. Conventional treatments (drugs, traditional herbal medications, rehabilitation therapies, or acupuncture therapies without electrostimulation for stroke and urinary incontinence / electroacupuncture therapies other than the acupoints (CV2, CV3, CV4, CV6, SP1 and SP6) for stroke and urinary incontinence) are permitted.
  Interventions: Device: Sham electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture (EA) — The EA group will receive the verum therapies using the following procedures.
  1. Let the patient lie down on lateral decubitus.
  2. The practitioners install the same guide-tubes as Park sham needle on CV2, CV3, CV4, CV6 and bilateral points of SP11 and SP6.
  3. The verum acupunctures are inserted on each acupoint inside the installed guide-tube. (stainless steel, 0.25 mm in diameter and 4.0 mm in length, Dong Bang Acupuncture Inc., Republic of Korea)
  4. After de qi response is elicited, the electrical stimulation is presented for 20 minutes by middle frequency (30 Hz). (STN-111, Stratek, Republic of Korea)
  5. The practitioner should have at least 1-year clinical experiences.
  The procedure will be repeated 10 times (once a session) within 21 days.
  Other Names: STN-111, Stratek, Republic of Korea
  Arms: Electroacupuncture (EA) group
Device: Sham electroacupuncture — 1. Let the patient lie down on lateral decubitus.
  2. The practitioners install the same guide-tubes as Park sham needle on CV2, CV3, CV4, and CV6 unilaterally & SP11 and SP6 bilaterally.
  3. The non-penetrating sham acupunctures are implemented on each acupoint inside the installed guide-tube.
  4. The electrical stimulation is presented for 20 minutes by middle frequency (30 Hz), (STN-111, Stratek, Republic of Korea) even though the electrical stimulation is not delivered through the skin because the needles are not penetrated through the skin.
  5. The practitioner should have at least 1-year clinical experiences.
  The procedure will be repeated 10 times (once a session) within 21 days.
  Other Names: Park sham device
  Arms: Park sham (PS) group

SUMMARY:
This pilot protocol is aimed to evaluate the effectiveness and safety of electroacupuncture therapy for the post-stroke patients with urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged over 19 years old
2. Patients diagnosed with stroke (cerebral hemorrhage or infarction) by the examination of computed tomography or magnetic resonance imaging methods within 2 years
3. Twice or more of urination with 3 to 4 points of PPIUS* at baseline OR 13 points or more of K-IPSS*
4. Any volunteers who signed the informed consent forms

Exclusion Criteria: We will exclude any patients with

1. Once or more of post-voiding residual > 200 ml per day
2. Clinically significant stress urinary incontinence diagnosed based on cough induction test or investigator's decision
3. Recurrent urinary tract infection defined as 4 or more treatments for urinary tract infection for the recent 1 year
4. Cognitive impairment with less than 23 points of MMSE-K* examination
5. Acute or chronic lower urinary tract infection examined by urine culture
6. Urinary incontinence diagnosed before the stroke occurred and the symptoms have continued until now based on medical history
7. Any severe diseases in lower urinary tract based on medical history and screening examination
8. Coagulation disorders based on medical history
9. Peripheral arterial diseases, which resulted in taking medical or surgical procedures to treat them based on medical history
10. Psychiatric diseases based on medical history
11. Fear of acupuncture based on questionnaire test
12. Pregnancy based on urine test
13. Any other inappropriate reasons on which the primary or sub investigators do not let the patients participate in the trial

    * Abbreviations PPIUS; Patient Perception of Intensity of Urgency Scale K-IPSS; The Korean version of International Prostate Symptom Scale MMSE-K; The Korean version of Mini-Mental State Examination

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Total Urgency and Frequency Score (TUFS) | at least 15 days (at most 21 days) (at baseline and the end of the treatment)
  The patients will be asked to fill the scale about their perception of urgency intensity (24 hours before the 1st session and after the last session, respectively) by themselves. They have to record every time of urination and select one of the 5 levels in perception of urgency intensity (0=No urgency, 1=Mild urgency, 2=Moderate urgency, 3=Severe urgency, 4= urgency incontinence) for 24 hours at baseline and the end of the treatment, respectively.

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire for Urinary Incontinence Short Form (ICIQ-UI-SF) | at least 15 days (at most 21 days) (at baseline and the end of the treatment)
The Korean version of International Prostate Symptom Scale (K-IPSS) | at least 15 days (at most 21 days) (at baseline and the end of the treatment)
The Lower urinary track system Outcome Score (LOS) | at least 15 days (at most 21 days) (at baseline and the end of the treatment)
Adverse events report | intraoperative

OTHER OUTCOMES:
Blinding Index (BI) | 21 days
  Patients will be asked to answer which arm they think they belonged to, assessing that the blinding succeed or not.

CONTACTS AND LOCATIONS:
Overall Officials: Euiju Lee, Ph.D., Principal Investigator — Kyunghee University
Locations (2):
- South Korea (2):
  - Wonkwang University Gwangju Medical Center, Gwangju
  - Kyung Hee University Korean Medicine Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Currie CT. Urinary incontinence after stroke. Br Med J (Clin Res Ed). 1986 Nov 22;293(6558):1322-3. doi: 10.1136/bmj.293.6558.1322-a. No abstract available. PMID 3790967
- [Background] Gelber DA, Good DC, Laven LJ, Verhulst SJ. Causes of urinary incontinence after acute hemispheric stroke. Stroke. 1993 Mar;24(3):378-82. doi: 10.1161/01.str.24.3.378. PMID 8446973
- [Background] Brittain KR, Perry SI, Peet SM, Shaw C, Dallosso H, Assassa RP, Williams K, Jagger C, Potter JF, Castleden CM. Prevalence and impact of urinary symptoms among community-dwelling stroke survivors. Stroke. 2000 Apr;31(4):886-91. doi: 10.1161/01.str.31.4.886. PMID 10753993
- [Background] Garrett VE, Scott JA, Costich J, Aubrey DL, Gross J. Bladder emptying assessment in stroke patients. Arch Phys Med Rehabil. 1989 Jan;70(1):41-3. PMID 2916918
- [Background] Mizrahi EH, Waitzman A, Arad M, Blumstein T, Adunksy A. Bladder management and the functional outcome of elderly ischemic stroke patients. Arch Gerontol Geriatr. 2011 Sep-Oct;53(2):e125-8. doi: 10.1016/j.archger.2010.07.007. Epub 2010 Aug 12. PMID 20708280
- [Background] Mustonen S, Ala-Houhala IO, Tammela TL. Long-term renal dysfunction in patients with acute urinary retention. Scand J Urol Nephrol. 2001 Feb;35(1):44-8. doi: 10.1080/00365590151030804. PMID 11291687
- [Background] Curtis LA, Dolan TS, Cespedes RD. Acute urinary retention and urinary incontinence. Emerg Med Clin North Am. 2001 Aug;19(3):591-619. doi: 10.1016/s0733-8627(05)70205-4. PMID 11554277
- [Background] Tibaek S, Gard G, Jensen R. Pelvic floor muscle training is effective in women with urinary incontinence after stroke: a randomised, controlled and blinded study. Neurourol Urodyn. 2005;24(4):348-57. doi: 10.1002/nau.20134. PMID 15791633
- [Background] Herr-Wilbert IS, Imhof L, Hund-Georgiadis M, Wilbert DM. Assessment-guided therapy of urinary incontinence after stroke. Rehabil Nurs. 2010 Nov-Dec;35(6):248-53. doi: 10.1002/j.2048-7940.2010.tb00055.x. PMID 21140719
- [Background] Tong Y, Jia Q, Sun Y, Hou Z, Wang Y. Acupuncture in the treatment of diabetic bladder dysfunction. J Altern Complement Med. 2009 Aug;15(8):905-9. doi: 10.1089/acm.2009.0062. PMID 19678782
- [Background] Mehdi Z, Birns J, Bhalla A. Post-stroke urinary incontinence. Int J Clin Pract. 2013 Nov;67(11):1128-37. doi: 10.1111/ijcp.12183. Epub 2013 Jul 8. PMID 23834208
- [Background] van Kerrebroeck P, Chapple C, Drogendijk T, Klaver M, Sokol R, Speakman M, Traudtner K, Drake MJ; NEPTUNE Study Group. Combination therapy with solifenacin and tamsulosin oral controlled absorption system in a single tablet for lower urinary tract symptoms in men: efficacy and safety results from the randomised controlled NEPTUNE trial. Eur Urol. 2013 Dec;64(6):1003-12. doi: 10.1016/j.eururo.2013.07.034. Epub 2013 Aug 3. PMID 23932438
- [Background] Chapple CR, Drake MJ, Van Kerrebroeck P, Cardozo L, Drogendijk T, Klaver M, Van Charldorp K, Hakimi Z, Compion G. Total urgency and frequency score as a measure of urgency and frequency in overactive bladder and storage lower urinary tract symptoms. BJU Int. 2014 May;113(5):696-703. doi: 10.1111/bju.12555. Epub 2014 Feb 20. PMID 24712917
- [Background] Abrams P, Avery K, Gardener N, Donovan J; ICIQ Advisory Board. The International Consultation on Incontinence Modular Questionnaire: www.iciq.net. J Urol. 2006 Mar;175(3 Pt 1):1063-6; discussion 1066. doi: 10.1016/S0022-5347(05)00348-4. PMID 16469618
- [Background] Hajebrahimi S, Nourizadeh D, Hamedani R, Pezeshki MZ. Validity and reliability of the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form and its correlation with urodynamic findings. Urol J. 2012 Fall;9(4):685-90. PMID 23235974
- [Background] Kang SG, Park CH, Kim DK, Park JK, Hong SJ, Chung BH, Kim CS, Lee KS, Kim JC, Lee JG. Long-term outcome of tamsulosin for patients with lower urinary tract symptoms according to the treatment response defined by lower urinary tract symptom outcomes score. Int J Clin Pract. 2011 Jun;65(6):691-7. doi: 10.1111/j.1742-1241.2011.02667.x. PMID 21564443
- [Background] Bang H, Ni L, Davis CE. Assessment of blinding in clinical trials. Control Clin Trials. 2004 Apr;25(2):143-56. doi: 10.1016/j.cct.2003.10.016. PMID 15020033